CLINICAL TRIAL: NCT06561750
Title: The Effect of Aspalathus Linearis on Muscle Soreness and Post-exercise Recovery in Young, Physically Inactive Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Daniel Afrifa, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CME2022/054
Record Dates: First submitted 2024-02-12; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Inflammation; Muscle Recovery; Muscle Soreness
Keywords: Aspalathus linearis; Rooibos
MeSH Terms: conditions — Inflammation; Myalgia

STUDY DESIGN:
Intervention Model Description: After undergoing a BIODEX exercise program to induce muscle soreness, participants will be randomised into 2 groups; the control and the aspalathus linearis groups. The Control group will be subjected to water while the aspalathus linearis group will be subjected to the rooibos tea
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rooibos (Experimental): Participants in the AG will consume the test drink (12 g per 1200 ml of pure green rooibos tea). Participants will be asked to return after 24, 48 and 72 hours of the exercise. During each visit, the baseline measurements, perceived muscle soreness and muscle recovery will be repeated.
  Interventions: Other: Rooibos tea
- Control (Placebo Comparator): Participants in the control group will be asked to drink 1200 ml of water since rooibos has a very unique taste
  Interventions: Other: Control

INTERVENTIONS:
Other: Rooibos tea — Participants will be subjected to 12 g of rooibos tea per 1200 ml of freshly boiled water
  Arms: Rooibos
Other: Control — Participants will be subjected to 12 g per 1200 ml of freshly boiled water which is equivalent to 6 cups of tea
  Arms: Control

SUMMARY:
Exercise has been found to exert beneficial effect on overall health. However, it also induces muscle damage at the same time. This then leads to muscle pain, temporary inflammation and reduced muscle function. These symptoms can persist for up to 72 hours after physical exertion and thus have a negative impact on a speedy recovery. Research has previously shown that antioxidants play an important role in muscle recovery after physical exertion. For example, antioxidants are known to have a positive effect on muscle damage and muscle soreness, and they also provide an anti-inflammatory effect. An important group of antioxidants are the flavonoids, which are abundantly present in rooibos (aspalathus linearis) tea. Previous research has shown that rooibos tea has a performance-enhancing effect during physical exertion. Despite these positive findings during physical exertion, the effect of rooibos tea on muscle recovery is not yet well known. Moreover, the effects of antioxidants during and after physical exertion have almost only been studied in men. Therefore, the current study will investigate the effects of rooibos tea on inflammation, muscle damage and muscle pain in a female population, and whether the muscle recovery capacity can ultimately be accelerated.

DETAILED DESCRIPTION:
On volunteers initial visit to the lab, they will be screened to assess their inclusion using the inclusion and exclusion criteria. Those who qualify for the study will be informed of the detailed procedures of the study. If they still decide to participate, they will be asked to read and sign the informed consent form. They will be asked to avoid taking NSAIDS during the course of the study. Participants will also be asked to refrain from the consumption of flavonoid-rich foods, drinks and supplements for 7 days prior to the test day. During the second visit (test day), baseline data such as body composition, anthropometrical variables, inflammatory markers (creatine kinase, TNF-α, IL-1 and IL-6), perceived muscle soreness and recover, and the quadriceps muscle functioning will be measured. The test will be done in the morning between 8:00 and 12:00 noon. To standardize the metabolic state of the participant during the testing sessions they will not be required to eat for at least two hours before testing. Moreover, participants will be required not to take caffeinated drinks and alcohol at least 12 hours before testing and not do any vigorous activities that have a rating of perceived exertion (RPE) more than (>) 12 on the Borg scale or any unusual exercise at least 24 hours before testing.

Participants will perform an 8 min warm-up of brisk walking on a treadmill (4-7 kph). They will then be subjected to the BIODEX exercise protocol. The protocol is composed of two exercise bouts (A and B), each of which comprises of 15 series of 12 maximum intermittent knee extensions conducted using the right leg on an isokinetic dynamometer with a 60 min break in between. During the 60 min break, the participants will cycle at 100 W on a bicycle ergometer (Monark) for 15 min in between bouts A and B, and then they rested in a semi-supine position for the next 45 min until bout B began. After completion of the exercise protocol, each participant will be asked to step down a total of four times from a bench 30.45 cm (1 ft.) high, alternating the leading leg between attempts to have each leg lead twice to assess the perceived muscle soreness using a 100-point visual analogue scale (VAS).

Participants will then be randomised into two (2) groups; the Aspalathus linearis group (AG) and the control group (CG). Participants will be asked to return after 24, 48 and 72 hours of the exercise. During each visit, the baseline measurements, perceived muscle soreness and muscle recovery will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Aged between 18-30 years
* Must not engage regularly in more than 2 organized resistance training session per week or more than 5 h physical activity per week for the previous six months.
* Answer "NO" to the seven questions of the Physical Activity Readiness Questionnaire plus (PAR-Q+) (Appendix B).

Exclusion Criteria:

* Pregnant or lactating
* Medication or undesirable alcohol consumption (>2 drinks per day) and smoking
* Have any medical condition that can have a serious impact on their ability to exercise or report acute illness, chronic disease or any other medical problems during the health screening (Appendix A) session that did not necessarily exclude them from physical activity by the PAR-Q+
* Currently using or have used vitamin and/or antioxidant supplementation for the last 2 months.
* Has a history of clotting disorders and are currently on non-steroidal anti-inflammatory drugs or anti-coagulants

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Serum creatine kinase from Baseline to 72 hours | Baseline and 72 hours
  Blood samples will be collected at baseline and 72 hours
Change in perceived muscle soreness from Baseline to 72 hours | Baseline and 72 hours
  A 10 point analogue scale will be used to assess the muscle soreness. The ratings on the scale are 0 = "no soreness or pain", 2 = "mild annoying pain", 4 = "Nagging, uncomfortable troublesome pain", 6 = "Distressing, miserable pain", 8 = "Intense, dreadful pain", and 10 = "the worst possible, unbearable, excruciating pain"
Change in perceived muscle recovery from Baseline to 72 hours | Baseline and 72 hours
  The perceived exercise recovery will be assessed using the Perceived recovery status (PRS) scale. The PRS scale rates recovery from exercise from 1 to 10 with 1-3 representing poor recovery and anticipating poor performance, 4-6 consisting of moderate recovery and expecting normal performance, and 7-10 representing high recovery and expecting increased performance
Change in Tumor Necrosis Factor -alpha (TNF-α) from Baseline to 72 hours | Baseline and 72 hours
  Blood samples will be collected at Baseline and 72 hours
Change in interleukin-6 (IL-6) from Baseline to 72 hours | Baseline and 72 Hours
  Blood samples will be collected at Baseline and 72 hours

SECONDARY OUTCOMES:
Change in swelling at the quadriceps muscle from Baseline to 72 hours | Baseline and 72 hours
  Quadriceps muscle swelling will be assessed using the thigh circumference measurement. The thigh circumference measurement will be done using the tape measure and performed to the nearest tenth of a centimeter. Two measurements within two millimeters of each other will be completed and averaged at each time point
Change in quadriceps contractile muscle functioning from Baseline to 72 hours | Baseline and 72 hours
  Quadriceps contractile muscle functioning will be assessed using vertical jump test. Squat jumps will be executed with both hands clasped together firmly behind the back to minimize arm assistance for uniformity after warming up with 12 squat jumps of rising height. The participants will be told to keep their trunks as erect as they could

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Afrifa, Principal Investigator — Hasselt University (HasseltU)
Locations (1):
- Biomedical Research Institute, Hasselt University, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data (IPD) that will be published will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After collection of data, it will be available for a maximum of 5 years
Access Criteria: Information will be shared with editors of the journal with which the data will be published. Researchers and individuals who may need the data for academic purposes may have to contact the investigator, the Biomedical Research Institute, Hasselt University for permission.
URL: http://www.uhasselt.be/en/instituten-en/biomed-en

REFERENCES:
- [Background] Sousa M, Teixeira VH, Soares J. Dietary strategies to recover from exercise-induced muscle damage. Int J Food Sci Nutr. 2014 Mar;65(2):151-63. doi: 10.3109/09637486.2013.849662. Epub 2013 Nov 4. PMID 24180469
- [Background] Marnewick JL, Rautenbach F, Venter I, Neethling H, Blackhurst DM, Wolmarans P, Macharia M. Effects of rooibos (Aspalathus linearis) on oxidative stress and biochemical parameters in adults at risk for cardiovascular disease. J Ethnopharmacol. 2011 Jan 7;133(1):46-52. doi: 10.1016/j.jep.2010.08.061. Epub 2010 Sep 15. PMID 20833235
- [Background] Eijnde BO, Van Leemputte M, Brouns F, Van Der Vusse GJ, Labarque V, Ramaekers M, Van Schuylenberg R, Verbessem P, Wijnen H, Hespel P. No effects of oral ribose supplementation on repeated maximal exercise and de novo ATP resynthesis. J Appl Physiol (1985). 2001 Nov;91(5):2275-81. doi: 10.1152/jappl.2001.91.5.2275. PMID 11641371
- [Background] Laurent CM, Green JM, Bishop PA, Sjokvist J, Schumacker RE, Richardson MT, Curtner-Smith M. A practical approach to monitoring recovery: development of a perceived recovery status scale. J Strength Cond Res. 2011 Mar;25(3):620-8. doi: 10.1519/JSC.0b013e3181c69ec6. PMID 20581704